CLINICAL TRIAL: NCT00069199
Title: Optical Coherence Tomography Comparative Study
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030294; 03-EI-0294
Record Dates: First submitted 2003-09-17; First posted 2003-09-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Retinal Disease; Healthy
Keywords: Reproducibility; Macular Edema; OCT2; OCT3; Retina
MeSH Terms: conditions — Retinal Diseases; Macular Edema

SUMMARY:
This study, conducted at the NIH Clinical Center and the University of Wisconsin University, will compare measurements obtained using older and newer models of a machine called an optical coherence tomography (OCT) scanner. This instrument uses a beam of light to measure the thickness of the retina, the light-sensitive inner lining of the back of the eye. OCT measurements will be done in multicenter clinical trials of new treatments for disorders that cause vision loss, such as macular edema. Because some centers in these studies will use the older OCT model and some the newer one, it is necessary to determine whether the two models give comparable results.

People 18 years of age and older in the following categories may be eligible for this study:

* People with diabetes, with or without macular edema;
* People with other retinal disease, such as uveitis or vein occlusion in the retina;
* People with no history of eye disease who have a normal retina.

Participants will have the following tests and procedures:

* Eye examination to assess vision and eye pressure and to evaluate the retina. The pupils are dilated with drops for this examination.
* Stereoscopic color fundus photography to examine the back of the eye. Eye drops are used to enlarge the size of the pupils to allow for a through examination and photographs of the eye using a special camera that flashes a bright light into the eye.
* OCT to measure retinal thickness. For this procedure, the subject sits in front of a small screen and looks at a target in the center of the screen while a dim red light moves across the subject's retina. This test is done first with one model of the OCT scanner, then the other. Finally, the test is repeated in both eyes with whichever model was used first.

Patients who are being treated for macular edema will repeat the same tests at their 3-month visits.

DETAILED DESCRIPTION:
The use of the Optical Coherence Tomography (OCT) has increased markedly over the recent years for clinical research. It is a promising new method for imaging the retina, measuring its thickness, and displaying some features of this structure. It is useful in assessing several eye diseases, including macular edema from various causes and abnormalities of the vitreoretinal interface. There is a broad clinical consensus that OCT is superior to stereoscopic color fundus photography, fluorescein angiography, and clinical biomicroscopic examination in measuring retinal thickness and is capable of documenting fairly small changes in thickness. OCT is becoming an important part of clinical trials of new treatments for macular edema. A number of models of the OCT device are commercially available, models 1, 2, and 3. A number of models of OCT have been used in clinical centers involved in such clinical research. Comparisons of these models 2 and 3 as well as the reproducibility of these measurements have not been conducted. The main research questions to be answered in this protocol are the following, in patients with normal retina, diabetic macular edema, macular edema from other causes, or other vitreoretinal abnormalities:

1. Is the standard deviation of the differences of sequential measurements of retinal thickness in normal retinas using OCT 3 similar to those measured with the OCT 2?
2. Are there systematic differences between thickness measurements using OCT 2 and OCT 3 in the same eyes?
3. Are there differences in the ability of each machine to image abnormalities within the vitreoretinal interface?

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient must understand and sign the informed consent.
2. Patient must be at least 18 years of age.
3. Pupillary dilation to at least 6 mm must be possible.
4. Ocular media must be sufficiently clear to allow for quality images.

EXCLUSION CRITERIA:

1. Any condition such as corneal opacifiation that precludes adequate slit lamp examination and photography of the fundus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hee MR, Puliafito CA, Duker JS, Reichel E, Coker JG, Wilkins JR, Schuman JS, Swanson EA, Fujimoto JG. Topography of diabetic macular edema with optical coherence tomography. Ophthalmology. 1998 Feb;105(2):360-70. doi: 10.1016/s0161-6420(98)93601-6. PMID 9479300
- [Background] Strom C, Sander B, Larsen N, Larsen M, Lund-Andersen H. Diabetic macular edema assessed with optical coherence tomography and stereo fundus photography. Invest Ophthalmol Vis Sci. 2002 Jan;43(1):241-5. PMID 11773037
- [Background] Otani T, Kishi S, Maruyama Y. Patterns of diabetic macular edema with optical coherence tomography. Am J Ophthalmol. 1999 Jun;127(6):688-93. doi: 10.1016/s0002-9394(99)00033-1. PMID 10372879